CLINICAL TRIAL: NCT02969837
Title: Open-label, Single-arm, Phase 2 Study of Initial Treatment With Elotuzumab, Carfilzomib (Kyprolis), Lenalidomide (Revlimid) and Low Dose Dexamethasone (E-KRd) in Newly Diagnosed, Multiple Myeloma Requiring Systemic Chemotherapy
Brief Title: Study of Initial Treatment With Elotuzumab, Carfilzomib, Lenalidomide and Dexamethasone in Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Bristol-Myers Squibb (Industry); Amgen (Industry); Multiple Myeloma Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB16-1138
Record Dates: First submitted 2016-11-14; First posted 2016-11-21 (Estimated); Results first posted 2025-09-10 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Elotuzumab; Carfilzomib (Kyprolis); Lenalidomide (Revlimid); Dexamethasone (E-KRd)
MeSH Terms: conditions — Multiple Myeloma | interventions — elotuzumab; carfilzomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: All participants will receive E-KRd regimen (elotuzumab, carfilzomib, lenalidomide, and dexamethasone) for up to 12 Cycles.
  After Cycle 12, participants that are MRD negative will move to E-Rd (elotuzumab, carfilzomib, lenalidomide, and dexamethasone) maintenance regimen and continue until disease progression. Participants that are MRD positive will continue to receive E-KRd regimen for an additional 6 cycles followed by E-Rd maintenance regimen and continue until disease progression
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Elo-KRd regimen (Experimental): Subjects will be tested for Minimal Residual Disease (MRD) by Next Generation Sequencing (NGS) and flow cytometry after cycles 8 and 12. A treatment decision was made after cycle 12 based on these results. There are three outcomes based on the IFM trial (Avet-Loiseau et al., 2015): 1) if the subject is MRD-negative by NGS after cycle 8 and 12, the subject went on E-Rd maintenance until disease progression. 2) If the subject is MRD-positive after cycle 8 but MRD-negative after cycle 12, 6 more cycles of E-KRd was given and at the end of 18 cycles, the subject went on E-Rd maintenance until disease progression. 3) Finally, if the subject is MRD-positive at both instances, 12 additional cycles of E-KRd was given and at the end of 24 cycles total, the subject went on E-Rd maintenance until disease progression.
  Interventions: Drug: Elotuzumab; Drug: Carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Elotuzumab — Elotuzumab will be given on Cycles 1-2 on days 1, 8, 15, 22, Cycles 3 and Beyond on days 1 and 15
  Other Names: Empliciti
Drug: Carfilzomib — Carfilzomib will be given on Day 1 and 8 of Cycle 1, Days 1, 8, and 15 of Cycles 2-8, and Days 1 and 15 of Cycles 9 and beyond
  Other Names: Kryprolis
Drug: Lenalidomide — Lenalidomide will be given on days 1-21 for all cycles.
  Other Names: Revlimid
Drug: Dexamethasone — Dexamethasone will be given as follows:
  Cycle 1 and 2: Days 1, 2, 8, 9, 15, 16, and 22 Cycles 3 and Beyond: Days 1, 8, 15, and 22

SUMMARY:
This study was a multi-center, open-label, single-arm, Phase 2 study where newly diagnosed Multiple Myeloma requiring systemic chemotherapy will be eligible for enrollment. A total of 46 subjects were enrolled. The primary end point was the rate of stringent complete response (sCR) and/or MRD-negativity (10-5) after C8 Elo-KRd. Secondary end points included safety, rate of response, MRD status, PFS, and overall survival (OS).

DETAILED DESCRIPTION:
Primary Objective

• The primary efficacy endpoint will be the rate of sCR and/or the rate of negative MRD by next generation gene sequencing (NGS) by clonoSIGHT (Adaptive Biotechnologies) at the end of 8 cycles among non-transplant candidates and transplant candidates who agreed to defer transplant

Secondary Objectives

* To evaluate the safety and tolerability of elotuzumab in combination with KRd, when administered to subjects with newly diagnosed multiple myeloma.
* To determine the rate of MRD by next generation gene sequencing (NGS) by clonoSIGHT (Adaptive Biotechnologies) and by multi-color flow cytometry (MFC) at the end of Cycle 4, 8,and 12 for all subjects, and end of C18 (for subjects who are MRD+ at the end of C8 but MRD- at the end of C12 only), 24 months after C1D1, and yearly after that.
* To estimate time to event, including duration of response (DOR), progression-free survival (PFS), time to progression (TTP), and overall survival (OS).

Exploratory Objectives

* GEP, proteomics, and gene sequencing to evaluate the correlation between treatment outcome and pre-treatment subject profile.
* Immunologic correlative studies including FcγRIIIa V genotype.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be eligible to enroll in this study. No enrollment waivers will be granted.

  1. Newly diagnosed, previously untreated myeloma requiring systemic chemotherapy

     a. Prior treatment of hypercalcemia or spinal cord compression or active and/or aggressively progressing myeloma with corticosteroids and/or lenalidomide and/or bortezomib/PI-based regimens does not disqualify the subject (the corticosteroid treatment dose should not exceed the equivalent of 160 mg of dexamethasone in a 4 week period or not more than 1 cycle of lenalidomide and/or PI-based therapy)
  2. Both transplant and non-transplant candidates are eligible.
  3. Diagnosis of symptomatic multiple myeloma as per current IMWG uniform criteria prior to initial treatment
  4. Monoclonal plasma cells in the BM 10% or presence of a biopsy-proven plasmacytoma
  5. Measurable disease, prior to initial treatment as indicated by one or more of the following:

     1. Serum M-protein ≥ 1 g/dL
     2. Urine M-protein ≥ 200 mg/24 hours
     3. If serum protein electrophoresis is felt to be unreliable for routine M-protein measurement, then quantitative immunoglobulin levels are acceptable (≥ 1 g/dL)
     4. Involved serum free light chains ≥ 10 mg/dL provided that free light chain ratio is abnormal
  6. Screening laboratory values must meet the following criteria and should be obtained within 21 days prior to enrollment WBC ≥ 2000/µL Platelets ≥ 75 x103/µL ANC >1000/µL Hemoglobin > 8.0 g/dL Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 50 mL/min

     1. Use the Cockcroft-Gault formula below):

        o Female CrCl = (140 - age in years) x weight in kg x 0.85
        * 72 x serum creatinine in mg/dL

          o Male CrCl = (140 - age in years) x weight in kg x 1.00
        * 72 x serum creatinine in mg/dL
     2. Alternatively to Cockcroft-Gault formula of CrCl, 24hr urine CrCl can be used AST/ALT ≤ 3 x ULN Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL) or ≤ 2 x ULN if lenalidomide is being prescribed.
  7. Males and females ≥ 18 years of age
  8. ECOG performance status of 0-1
  9. Females of childbearing potential (FCBP) must have 2 negative pregnancy tests (sensitivity of at least 50 mIU/mL) prior to initiating lenalidomide. The first pregnancy test must be performed within 10-14 days before and the second pregnancy test must be performed within 24 hours before lenalidomide is prescribed for Cycle 1 (prescriptions must be filled within 7 days).
  10. FCBP must agree to use 2 reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) for at least 28 days before starting lenalidomide; 2) while participating in the study; and 3) for at least 28 days after discontinuation from the study.
  11. Male subjects must agree to use a latex condom during sexual contact with females of childbearing potential while participating in the study and for at least 28 days following discontinuation from the study even if he has undergone a successful vasectomy.
  12. All study participants in the US must be consented to and registered into the mandatory Revlimid REMS program and be willing and able to comply with the requirements of Revlimid REMS.
  13. Voluntary written informed consent

Exclusion Criteria:

* Subjects meeting any of the following exclusion criteria are not eligible to enroll in this study. No enrollment waivers will be granted.

  1. Non-secretory or hyposecretory multiple myeloma, prior to initial treatment defined as <1.0 g/dL M-protein in serum, <200 mg/24 hr urine M-protein, and no measurable disease as per IMWG by Freelite.
  2. POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
  3. Geriatric assessment score of ≥2 as defined by Palumbo et al.
  4. Known or suspected Amyloidosis
  5. Plasma cell leukemia
  6. Within 4 weeks since any plasmapheresis
  7. Within 3 weeks of any corticosteroids except per inclusion criteria #2
  8. Waldenström's macroglobulinemia or IgM myeloma
  9. Participation in an investigational therapeutic study within 3 weeks or within 5 drug half-lives (t1/2) prior to first dose, whichever time is greater
  10. Subjects not able to tolerate elotuzumab, lenalidomide, carfilzomib, or dexamethasone
  11. Peripheral neuropathy ≥ Grade 2 at screening
  12. Prior CVA with persistent neurological deficit
  13. Diarrhea > Grade 1 in the absence of antidiarrheals
  14. CNS involvement
  15. Corrected calcium ≥ 11.5 mg/dL within 2 weeks of randomization
  16. Pregnant or lactating females
  17. Radiotherapy within 14 days before randomization. Seven days may be considered if to single area
  18. Major surgery within 3 weeks prior to first dose
  19. Subject has clinically significant cardiac disease, including:

      * myocardial infarction within 1 year before Cycle 1 Day 1, or an unstable or uncontrolled disease/condition related to or affecting cardiac function (eg, unstable angina, congestive heart failure, New York Heart Association Class III-IV
      * uncontrolled cardiac arrhythmia (NCI CTCAE Version 4 Grade 2:2) or clinically significant ECG abnormalities
      * screening 12-lead ECG showing a baseline QT interval as corrected by Fridericia's formula (QTcF) >470 msec
  20. Uncontrolled HTN 14 days prior to enrollment
  21. Prior or concurrent deep vein thrombosis or pulmonary embolism
  22. Rate-corrected QT interval of electrocardiograph (QTc) > 470 msec on a 12-lead ECG during screening
  23. Uncontrolled hypertension (defined as average systolic blood pressure ≥140 or average diastolic blood pressure ≥90, with blood pressure measured ≥3 times in the two weeks prior to enrollment ) or diabetes
  24. Acute infection requiring systemic antibiotics, antivirals, or antifungals within two weeks prior to first dose
  25. Active infection
  26. Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Subjects who are seropositive because of hepatitis B virus vaccine are eligible.
  27. Non-hematologic malignancy or non-myeloma hematologic malignancy within the past 3 years except a) adequately treated basal cell, squamous cell skin cancer, thyroid cancer, carcinoma in situ of the cervix, or prostate cancer < Gleason Grade 6 with stable prostate specific antigen levels or cancer considered cured by surgical resection alone
  28. Any clinically significant medical disease or condition that, in the Treating Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2025-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Jakubowiak, MD, Principal Investigator — University of Chicago
Locations (3):
- United States (3):
  - University of Chicago, Chicago, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan

REFERENCES:
- [Derived] Derman BA, Kansagra A, Zonder J, Stefka AT, Grinblatt DL, Anderson LD Jr, Gurbuxani S, Narula S, Rayani S, Major A, Kin A, Jiang K, Karrison T, Jasielec J, Jakubowiak AJ. Elotuzumab and Weekly Carfilzomib, Lenalidomide, and Dexamethasone in Patients With Newly Diagnosed Multiple Myeloma Without Transplant Intent: A Phase 2 Measurable Residual Disease-Adapted Study. JAMA Oncol. 2022 Sep 1;8(9):1278-1286. doi: 10.1001/jamaoncol.2022.2424. PMID 35862034

RESULTS

PARTICIPANT FLOW:
Groups:
- Elo-KRd Regimen: Subjects will be tested for Minimal Residual Disease (MRD) by Next Generation Sequencing (NGS) and flow cytometry after cycles 8 and 12. A treatment decision was made after cycle 12 based on these results. There are three outcomes based on the IFM trial (Avet-Loiseau et al., 2015): 1) if the subject is MRD-negative by NGS after cycle 8 and 12, the subject went on E-Rd maintenance until disease progression. 2) If the subject is MRD-positive after cycle 8 but MRD-negative after cycle 12, 6 more cycles of E-KRd was given and at the end of 18 cycles, the subject went on E-Rd maintenance until disease progression. 3) Finally, if the subject is MRD-positive at both instances, 12 additional cycles of E-KRd was given and at the end of 24 cycles total, the subject went on E-Rd maintenance until disease progression.
  Elotuzumab: Elotuzumab will be given on Cycles 1-2 on days 1, 8, 15, 22, Cycles 3 and Beyond on days 1 and 15
  Carfilzomib: Carfilzomib will be given on Day 1 and 8 of Cycle 1, Days 1, 8, and 15 of Cycles 2-8, and Days 1 and 15 of Cycles 9 and beyond
  Lenalidomide: Lenalidomide will be given on days 1-21 for all cycles.
  Dexamethasone: Dexamethasone will be given as follows:
  Cycle 1 and 2: Days 1, 2, 8, 9, 15, 16, and 22 Cycles 3 and Beyond: Days 1, 8, 15, and 22
Period: Overall Study
Arm/Group | Elo-KRd Regimen
Started | 46
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Elo-KRd Regimen
Number analyzed (Participants) | 46
Age, Continuous [Median (Full Range); unit: years] | 62 [43 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 32
  More than one race | 3
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Stringent Complete Response (sCR)
Description: Response will be determined according to the International Myeloma Working Group (IMWG) response criteria for multiple myeloma.
  sCR is defined as CR plus :
  * normal FLC ratio and
  * absence of clonal cells in bone marrow by immunohistochemistry or 2 - 4 color flow cytometry
  CR is defined as below :
  * Negative immunofixation on the serum and urine and
  * disappearance of any soft tissue plasmacytomas and
  * < 5% plasma cells in bone marrow.
  * In subjects with only FLC disease, a normal FLC ratio of 0.26-1.65 is required.
Time Frame: Landmark evaluations were performed after cycles 4, 8, 12, 18 and 24 (that is, 4, 8, 12, 18 and 24 months)
Population: One censored because of autologous stem cell transplant cycle 8 without progression
Measure: Count of Participants; unit: Participants
Arm/Group | Elo-KRd Regimen
Number analyzed (Participants) | 45
Participants | 17

2. Primary Outcome: Number of Participants With MRD-negativity (10^-5) After C8 Elo-KRd
Description: Subjects will be tested for Minimal Residual Disease (MRD) by Next Generation Sequencing (NGS) and flow cytometry after cycle 8.
  The flow cytometry analysis procedure used to determine MRD is performed on a NAVIOS FLOW CYTOMETER SYSTEM manufactured by BECKMAN COULTER, INC., using a laboratory developed assay.
  The Premarket Notification 510(k) (Number K130373) for the device can be found using the following link.
  https://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfpmn/pmn.cfm?ID=K130373.
Time Frame: Landmark evaluations were performed after cycle 8
Population: One censored because of autologous stem cell transplant cycle 8 without progression
Measure: Count of Participants; unit: Participants
Arm/Group | Elo-KRd Regimen
Number analyzed (Participants) | 45
Participants | 26

3. Primary Outcome: The Number of Participants With Stringent Complete Response (sCR) and/or MRD Negative (10^-5) by NGS
Description: Response will be determined according to the International Myeloma Working Group (IMWG) response criteria for multiple myeloma.
  sCR is defined as CR plus :
  * normal FLC ratio and
  * absence of clonal cells in bone marrow by immunohistochemistry or 2 - 4 color flow cytometry
  CR is defined as below :
  * Negative immunofixation on the serum and urine and
  * disappearance of any soft tissue plasmacytomas and
  * < 5% plasma cells in bone marrow.
  * In subjects with only FLC disease, a normal FLC ratio of 0.26-1.65 is required.
  Subjects will be tested for Minimal Residual Disease (MRD) by Next Generation Sequencing (NGS) and flow cytometry after cycles 4,8,12,18 and 24.
  The flow cytometry analysis procedure used to determine MRD is performed on a NAVIOS FLOW CYTOMETER SYSTEM manufactured by BECKMAN COULTER, INC., using a laboratory developed assay.
Time Frame: Landmark evaluations were performed after cycles 4, 8, 12, 18 and 24 (that is, 4, 8, 12, 18 and 24 months)
Population: One censored because of autologous stem cell transplant cycle 8 without progression
Measure: Count of Participants; unit: Participants
Arm/Group | Elo-KRd Regimen
Number analyzed (Participants) | 45
Participants | 26

4. Secondary Outcome: Number of Participants With Adverse Events of Elotuzumab in Combination With KRd
Description: AEs were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (version 4.0)
Time Frame: AEs were recorded from the day of signed consent through 30 days after the last does of Elo-KRd or initiation of new therapy, an average of 2 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Elo-KRd Regimen
Number analyzed (Participants) | 46
Participants
  Anemia | 11
  Neutropenia | 9
  Thrombocytopenia | 8
  Lymphopenia | 4
  Fatigue | 33
  Infection-Upper respiratory | 19
  Infection-Non-pulmonary | 22
  Infection-Lung | 7
  Infection-Bronchial | 2
  Diarrhea | 29
  Dyspnea | 20
  Peripheral neuropathy | 19
  Nausea | 16
  Hyperglycemia | 14
  Cardia events, any | 12
  Electrolyte imbalances, any | 12
  Hypertension | 11
  Rash | 7
  Thromboembolic events | 5
  Infusion reactions | 5
  Acute kidney injury | 5

5. Secondary Outcome: Duration of Response
Description: These events will be analyzed at differing points of time based on the individual subjects disease progression. It will be measured by the number of cycles of therapy.
Time Frame: Up to two years
Measure: Median (Full Range); unit: cycles of therapy
Arm/Group | Elo-KRd Regimen
Number analyzed (Participants) | 46
cycles of therapy | 23 [2 to 39]

6. Secondary Outcome: Median Progression Free Survival
Description: Progression free survival (PFS) was assessed based on time to disease progression or death (whichever occurred first) from the start of treatment.
Time Frame: up to two years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Elo-KRd Regimen
Number analyzed (Participants) | 46
months | NA [NA to NA] — Median PFS has not been reached due to insufficient number of participants with events.

7. Secondary Outcome: Median Overall Survival
Description: Overall survival (OS) was assessed based on time to disease progression or death (whichever occurred first) from the start of treatment.
Time Frame: up to two years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Elo-KRd Regimen
Number analyzed (Participants) | 46
months | NA [NA to NA] — Median OS has not been reached due to insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Elo-KRd Regimen
All-Cause Mortality (participants affected / at risk) | 8/46
Serious Adverse Events (participants affected / at risk) | 18/46
Other Adverse Events (participants affected / at risk) | 42/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Elo-KRd Regimen (N=46)
Acute kidney injury (Renal and urinary disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Bronchial infection (Infections and infestations) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Ejection fraction decreased (Investigations) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Fever (General disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infections and infestations - Other (Infections and infestations) | 1
Lung infection (Infections and infestations) | 5
Myocardial infraction (Cardiac disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Renal and urinary disorders - Other (Renal and urinary disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Elo-KRd Regimen (N=46)
Agitation (Psychiatric disorders) | 3
Alanine aminotransferase increased (Investigations) | 9
Anemia (Blood and lymphatic system disorders) | 7
Aspartate aminotransferase increased (Investigations) | 4
Atrial fibrillation (Cardiac disorders) | 3
Blurred vision (Eye disorders) | 4
Constipation (Gastrointestinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 21
Dizziness (Nervous system disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13
Edema limbs (General disorders) | 17
Fatigue (General disorders) | 29
Fever (General disorders) | 8
Hyperglycemia (Metabolism and nutrition disorders) | 11
Hypertension (Vascular disorders) | 7
Infusion related reaction (General disorders) | 4
Insomnia (Psychiatric disorders) | 13
Localized edema (General disorders) | 7
Lymphocyte count decreased (Investigations) | 3
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 7
Nausea (Gastrointestinal disorders) | 14
Neutrophil count decreased (Investigations) | 6
Paresthesia (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 17
Platelet count decreased (Investigations) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6
Skin and subcutaneous tissue disorders- Other (Skin and subcutaneous tissue disorders) | 5
Thromboembolic event (Vascular disorders) | 4
Tremor (Nervous system disorders) | 4
Upper respiratory infection (Infections and infestations) | 7
Vomiting (Gastrointestinal disorders) | 3
Weight gain (Investigations) | 5
White blood cell decreased (Investigations) | 10
Cardiac disorders - Other (Cardiac disorders) | 3
Chills (General disorders) | 3
Dysgeusia (Nervous system disorders) | 3
Flu like symptoms (General disorders) | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4
General disorders and administration site conditions-Other (General disorders) | 3
Headache (Nervous system disorders) | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 5
Hypotension (Vascular disorders) | 3
Mucositis oral (Gastrointestinal disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Sinusitis (Infections and infestations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/37/NCT02969837/Prot_SAP_000.pdf